CLINICAL TRIAL: NCT05112770
Title: AI for Allograft Diseases Diagnosis and Prognosis After Kidney Transplantation
Acronym: AI4ADAPT
Status: Withdrawn | Type: Observational
Why Stopped: 29 / 5 000 Abandoned research project
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210907
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Acute renal transplant rejection; Urinary concentrations of chemokines; Multiparametric models; Artificial intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Renal transplant patients whose medical follow-up is provided from 2004 to 2020 by the nephrology and adult renal transplantation department of the Necker hospital.

SUMMARY:
Kidney transplantation is the treatment of choice for patients with end stage renal disease. One of the major challenges is to better diagnose the attacks undergone by the kidney transplant in order to increase its longevity. Multiple attacks are caused by non-immune and immune mechanisms, first and foremost the acute rejection of the transplant.

Biopsy, an invasive method, remains the "Gold Standard" for diagnosing rejection and other pathologies affecting the kidney transplant.

The invasive nature of these biopsies limits their use and alternative biomarkers have been evaluated in order to diagnose kidney transplant pathologies in a non-invasive manner. It is in this context that the nephrology and renal transplantation department of the Necker hospital and Inserm U1151 have carried out several studies leading to the identification of the diagnostic and prognostic potential of acute rejection, by the determination of urinary concentrations of two chemokines, CXCL9 and CXCL10.

The most recent study conducted within these teams demonstrated that the diagnostic potential of urinary chemokines could be improved by taking into account standard clinicobiological parameters in multiparametric models.

The main objective of the study is to develop, train and validate artificial intelligence models including urinary chemokines, efficient, robust, explainable and interpretable for the diagnosis and non-invasive prognosis of acute renal transplant rejection, trained on a data set made up of clinical and biological parameters.

DETAILED DESCRIPTION:
Kidney transplantation is the treatment of choice for patients with end stage renal disease. One of the major challenges is to better diagnose the attacks undergone by the kidney transplant in order to increase its longevity. Multiple attacks are caused by non-immune and immune mechanisms, first and foremost the acute rejection of the transplant.

Biopsy, an invasive method, remains the "Gold Standard" for diagnosing rejection and other pathologies affecting the kidney transplant.

The invasive nature of these biopsies limits their use and alternative biomarkers have been evaluated in order to diagnose kidney transplant pathologies in a non-invasive manner. It is in this context that the nephrology and renal transplantation department of the Necker hospital and Inserm U1151 have carried out several studies leading to the identification of the diagnostic and prognostic potential of acute rejection, by the determination of urinary concentrations of two chemokines, CXCL9 and CXCL10.

The most recent study conducted within these teams demonstrated that the diagnostic potential of urinary chemokines could be improved by taking into account standard clinicobiological parameters in multiparametric models.

The main objective of the study is to develop, train and validate artificial intelligence models including urinary chemokines, efficient, robust, explainable and interpretable for the diagnosis and non-invasive prognosis of acute renal transplant rejection, trained on a data set made up of clinical and biological parameters.

For this, all the clinical parameters (demographic, medical history, characteristics of donors, immunosuppressive treatments, etc.) and biological (follow up of the usual biological parameters obtained as part of the routine care of transplant patients, urinary chemokines) of transplant patients followed in the nephrology and renal transplantation department of Necker hospital between 2004 and 2020, will be treated without a priori and by artificial intelligence methods.

ELIGIBILITY:
Inclusion Criteria:

* All renal transplant patients whose medical follow-up is provided by the nephrology and adult renal transplantation department of the Necker hospital between 2004 and 12/31/2020;
* Patient having signed a consent form for the storage, use and transfer of samples taken during treatment, for scientific research purposes;
* Patient not objecting to the processing of his personal data as part of the study.

Exclusion Criteria:

- A deceased patient who, during his lifetime, objected in writing to the processing of his data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All renal transplant patients whose medical follow-up is provided by the nephrology and adult renal transplantation department of the Necker hospital between 2004 and 12/31/2020.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic model accuracy | 3 years
  ROC (receiver operating characteristic) curves AUC (Area under the Curve)
Prognostic model accuracy | 3 years
  C-statistics

SECONDARY OUTCOMES:
Strenght of the models | 3 years
  Sensitivity analyses comparing the AUC values and the calibration of the models in various clinical scenarios.

CONTACTS AND LOCATIONS:
Overall Officials: Dani Anglicheau, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No